CLINICAL TRIAL: NCT01531114
Title: Prasugrel Or Ticagrelor In ST-Elevation Myocardial Infarction Patients With Diabetes Mellitus
Brief Title: PraSugrel vs TicagrElor in ST-Elevation Myocardial Infarction paTients With Diabetes Mellitus
Acronym: RESET 2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gennaro Sardella (Other)
Responsible Party: Sponsor-Investigator, Gennaro Sardella, Associate Professor in Cardiology, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESET 2D Trial
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: Diabetes mellitus; antiplatelet effect; prasugrel; ticagrelor; STEMI; Insulin
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus; Insulin Resistance | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel loading dose (Active Comparator): Patients will be randomized to this arm to receive loading dose of prasugrel
  Interventions: Drug: ticagrelor; Drug: prasugrel
- ticagrelor loading dose (No Intervention): Patients will be randomized to this arm to receive loading dose of ticagrelor

INTERVENTIONS:
Drug: ticagrelor — Patients will be randomized to this arm to receive loading dose of ticagrelor
  Arms: Prasugrel loading dose
Drug: prasugrel — Patients will be randomized to this arm to receive loading dose of prasugrel
  Arms: Prasugrel loading dose

SUMMARY:
Dual antiplatelet therapy is essential in patients following ST-Elevation myocardial infarction (STEMI) with percutaneous coronary intervention (PCI) and drug eluting stent implantation. Current guidelines recommend prasugrel and ticagrelor in patients with STEMI undergoing primary PPCI. We sought to investigate the superiority antiplatelet effect in terms of PR level of loading dose (LD) of Prasugrel (60 mg) versus LD of Ticagrelor (180 mg) in diabetic patients with STEMI undergoing primary PCI at 1 and 2 hours post drug administration. Secondary end-points will be: PR level measured at 6 and 12 hours post study drugs administrationin hospital. All consecutive diabetic patients with STEMI undergoing PPCI with stent implantation will be considered for PR assessment at 1-2-6-12 h after the drug LD administration. All patients must will be naïve for platelet P2Y12 receptor inhibition therapy. A subanalysis will be performed between two study groups according to insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* acute coronary syndrome
* patients underwent to primary PCI
* naïve for platelet P2Y12 receptor inhibition therapy

Exclusion Criteria:

* history of bleeding diathesis
* chronic oral anticoagulation treatment
* contraindications to antiplatelet therapy
* PCI or coronary artery bypass grafting (CABG) < 3 months
* hemodynamic instability
* platelet count < 100,000/μl
* hematocrit < 30%
* creatinine clearance < 25 ml/min
* Patients with a history of stroke
* contraindication for prasugrel administration
* patients weighing < 60 kg
* patients treated with morphine
* > 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the superiority antiplatelet effect in terms of PR level of loading dose (LD) of Prasugrel (60 mg) versus LD of Ticagrelor (180 mg) in diabetic patients with STEMI undergoing primary PCI at 2 hours post drug administration. | 1 and 2 hours

SECONDARY OUTCOMES:
PR level measured at 6 and 12 hours post study drugs administration. | in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Dept.of Cardiovascular Sciences,Policlinico Umberto I, Rome, Italy